CLINICAL TRIAL: NCT05730114
Title: Platelet Aggregation in Patients Treated With P2Y12 Inhibitors and V-A ECMO for Cardiac Arrest
Brief Title: Monitoring Antiplatelet Drugs in Cardiac Arrest Patients
Acronym: PLT-ECMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Matteo Pozzi, MD, University of Milano Bicocca
Other Study IDs: 3940
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Cardiac Arrest; Myocardial Infarction; Extracorporeal Membrane Oxygenation; Platelet Dysfunction
MeSH Terms: conditions — Heart Arrest; Myocardial Infarction | interventions — Platelet Aggregation Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- OHCA/ECMO: Patient resuscitated from Out of Hospital Cardiac Arrest from acute coronary syndrome and on VA-ECMO.
  Interventions: Drug: Antiplatelet Drug
- OHCA/nonECMO: Patient resuscitated from Out of Hospital Cardiac Arrest from acute coronary syndrome and without VA-ECMO.
  Interventions: Drug: Antiplatelet Drug
- nonOHCA/nonECMO: Patient with acute coronary syndrome without Out of Hospital Cardiac Arrest from acute coronary syndrome and without VA-ECMO.
  Interventions: Drug: Antiplatelet Drug

INTERVENTIONS:
Drug: Antiplatelet Drug — anti-P2Y12 oral agent administered during primary percutaneous coronary intervention.

SUMMARY:
Dual Antiplatelet Therapy (DAPT) with acetylsalicylic acid (ASA) and oral P2Y12 inhibitor (Clopidogrel, Ticagrelor or Prasugrel) is recommended in STEMI or NSTEMI patients undergoing primary Percutaneous Coronary Intervention (PCI). There is evidence for an increased risk of stent thrombosis after PCI despite administration of DAPT in patients resuscitated from a cardiac arrest with STEMI/NSTEMI who undergo primary PCI, in particular for those treated with hypothermia. Point of Care Aggregometry represents an emerging tool to measure platelet reactivity in patient treated with antiplatelets drugs. Among patients with Acute Coronary Syndrome (ACS), those requiring Veno-Arterial Extracorporeal Membrane Oxygenation (VA-ECMO) for refractory Cardiogenic Shock or Cardiac Arrest represent a growing population burdened by more profound metabolic, pharmacokinetic, hemostatic and physiological alterations due to increased clinical severity and ECMO itself. In addition, profound platelet inhibition can result in a higher risk of bleeding complication, since these patients have to be simultaneously anticoagulated with unfractioned heparin (UFH) and ECMO itself can cause coagulopathy. We aimed to perform an observational prospective cohort study to investigate platelet reactivity in a population of ACS patients with different clinical severity.

ELIGIBILITY:
Inclusion Criteria:

* Patients P2Y12 naive
* Suffering from Acute Coronary Syndrome needing primary percutaneous coronary intervention (PCI) and treated with oral antiP2Y12 drugs

Exclusion Criteria:

* Known liver or hematological disease
* Anticoagulant therapy
* Active bleeding needing blood transfusions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted to ICU for Acute Coronary Syndrome and treated with oral P2Y12 inhibitors during primary PCI.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
HRPR risk | 7 days
  Relative risk to develop High Residual Platelet Reactivity (HRPR) during the first seven days of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Gerardo dei Tintori, Monza, MB, Italy

IPD SHARING:
Plan to Share IPD: Undecided